CLINICAL TRIAL: NCT01340807
Title: A Comparison of External Mechanical Work Between Bionic and Conventional Prosthetic Feet in Transtibial Amputees During Functional Activities
Brief Title: A Comparison of External Mechanical Work Between Different Prosthetic Feet
Acronym: SEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Ronald Tolchin, DO, Miami VAHS
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8497.01; 01 (Other: Miami VAHS)
Record Dates: First submitted 2011-04-19; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-02

CONDITIONS: Traumatic Amputation of Lower Extremity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prosthetic Feet (Experimental): Randomized to 4 different prosthetic feet (SACH, SAFE, TALUX, and Proprio Foot)
  Interventions: Other: Specialized Functional Prosthetic Training

INTERVENTIONS:
Other: Specialized Functional Prosthetic Training — Each subject receives specialized functional prosthetic training
  Other Names: Proshetic Feet

SUMMARY:
Recent dysvascular and diabetic amputees as well as older, long-term traumatic amputees are at risk of functional decline, joint degeneration, skin breakdown and further limb loss due to the forces placed on the contralateral limb through prosthetic ambulation. If specialized prosthetic gait training and proper use of the appropriate prosthetic foot can decrease forces on the intact limb, the long term health and quality of life of veterans with amputations could be substantially improved. We will address two key questions:

Key Question 1: After receiving specialized gait training and a new prosthetic socket, will subjects demonstrate differences in gait symmetry and external mechanical work between the bionic and conventional prosthetic feet, while performing various functional activities.

Key Question 2: Can external mechanical work be used as a clinically friendly measure to differentiate between prosthetic feet?

DETAILED DESCRIPTION:
The study examined the application of outcome measures to determine changes in function of unilateral transtibial amputees (TTAs) caused by specialized functional prosthetic training (training) and the use of four different prosthetic feet. Two self-report measures i.e. the Prosthetic Evaluation Questionnaire (PEQ-13) and Locomotor Capability Index (LCI-5), and three performance-based measures i.e. the Amputee Mobility Predictor (AMPPRO), Six-minute Walk Test (6MWT), and Step Activity Monitor (SAM) were utilized. Healthy unilateral Transtibial Amputees between the age of 40-65 will participate in the study. Subjects were tested at baseline, after receiving training with their existing prosthesis, and with the study socket and four prosthetic feet i.e. SACH, SAFE, Talux and PROPRIO FOOT over an 8-10 week period. Training was administered between testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or Females between the ages of 40 and 65. b. People with unilateral transtibial amputations for vascular reasons or from traumatic events.

  c. At the lowest level of function candidates will have the ability to use a prosthesis for ambulation on level surfaces at a fixed cadence.

  d. People with a diagnosis of diabetes mellitus and/or peripheral vascular disease leading to amputation or people who have been amputated as a result of trauma.

  e. People comfortably fitted with a prosthesis for a period of at least 6 months.

  f. Candidates who score within the range of 29 to 47 on the Amputee Mobility Predictor which would indicate that subjects achieved the minimum required score to be fitted with a prosthesis.

  g. Able to tolerate the testing protocol and would not fatigue at any time during testing.

  h. Men's shoe size should be between 7.5 (25 cm) and 12.5 (29 cm). i. Women's shoe size should be between 8.5 (25 cm) and 13.5 (29 cm).

Exclusion Criteria:

* People who weigh more than 255 pounds at baseline visit. People receiving renal dialysis b. People with severe cardiac or pulmonary disease limiting ability to exercise including angina or poorly controlled hypertension.

  c. People with neurological disorder such as or stroke that affecting ability to ambulate d. People with severe lower limb arthritis e. People with wound on non-amputated side f. People experiencing problems with prosthetic fit g. People with poor control of diabetes

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Symmetry in External Work | up to 12 weeks
  Work done by the intact and prosthetic limb

SECONDARY OUTCOMES:
Self Report and Performance Based Assessment Instruments | up to 12 weeks
  PEQ-13, LCI-5, AMPPRO, 6MWT, and SAM.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Tolchin, DO, Principal Investigator — Miami VAHS
Locations (1):
- Miami VAHS, Miami, Florida, United States